CLINICAL TRIAL: NCT05657444
Title: Intra-arterial Tenecteplase During First Thrombectomy Attempt for Acute Stroke (BRETIS-TNK II): a Prospective, Randomized, Adaptive Enrichment, Open-label, Blinded End Point, Multi-center Study
Brief Title: Intra-arterial Tenecteplase During First Thrombectomy Attempt for Acute Stroke (BRETIS-TNK II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Collaborators: Cerebrovascular Disease Collaboration & Innovation Alliance of Liaoning (Unknown)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Head of Neurology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2022) 168
Record Dates: First submitted 2022-12-02; First posted 2022-12-20 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNK group (Experimental)
  Interventions: Drug: Tenecteplase
- control group (No Intervention)

INTERVENTIONS:
Drug: Tenecteplase — intra-arterial tenecteplase during endovascular treatment
  Arms: TNK group

SUMMARY:
A recent pilot study suggests intra-arterial tenecteplase (TNK) during the first pass of endovascular treatment (EVT) seems safe, may increase first-pass reperfusion and good outcome in acute ischemic stroke (AIS) patients with large vessel occlusion (LVO).

The study aimed to determine the efficacy and safety of intra-arterial TNK administration during EVT in AIS-LVO patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Stroke patient with large vessel occlusion (internal carotid artery, M1 or M2 of middle cerebral artery, basilar artery, or intracranial segment of vertebral artery) who meets criteria for endovascular treatment within 24 hours of stroke onset;
* The modified Rankin Scale (mRS) score before onset ≤ 2;
* ASPECTS 6 or greater on CT
* Signed informed consent.

Exclusion Criteria:

* hemorrhagic stroke;
* Tandem occlusion;
* Coagulation disorders, systematic hemorrhagic tendency, thrombocytopenia (<100000/mm3);
* Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), elevated serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis;
* Severe uncontrolled hypertension (systolic blood pressure over 200mmHg or diastolic blood pressure over 110 mmHg);
* Patients with contraindication or allergic to any ingredient of drugs in our study;
* Pregnancy, or plan to get pregnant or during active lactation;
* Suspected septic embolus or infective endocarditis
* The estimated life expectancy is less than 6 months due to other serious diseases;
* Other conditions unsuitable for this clinical study as assessed by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
proportion of favorable outcome | Day 90
  Favorable outcome is defined as modified Rankin Scale (mRS) score of 0-2

SECONDARY OUTCOMES:
proportion of excellent outcome | Day 90
  Excellent outcome is defined as modified Rankin Scale (mRS) score of 0-1
proportion of successful reperfusion after the first-pass or final pass of endovascular treatment | immediately after the first-pass or final pass of endovascular treatment
  Successful reperfusion is defined as defined as modified Thrombolysis In Cerebral Infarction (mTICI) 2b-3
Distribution of modified Rankin Scale (mRS) | Day 90
  mRS scores range from 0 to 6:0, no symptoms, 1 = symptoms without clinically significant disability, 2 = slight disability, 3 = moderate disability, 4 = moderately severe disability, 5 = severe disability; and 6 = death.
Change in cerebral circulation time after intervention | immediately after endovascular treatment
occurrence rate of early neurological improvement | 24 (-6/+24) hours
  early neurological improvement was defined as a 4 point or greater decrease in NIHSS
change in National Institute of Health stroke scale (NIHSS) | 24 (-6/+24) hours
  NIHSS scores range 0-42, with higher scores indicating greater stroke severity
occurrence rate of the composite events of nonfatal stroke, nonfatal myocardial infarction, and other cardiovascular events | Day 90
occurrence rate of symptomatic intracranial hemorrhage | 24 (-6/+24) hours
  symptomatic intracranial hemorrhage is defined as an increase in the NIHSS score of ≥4 points as a result of the intracranial hemorrhage.
occurrence rate of parenchymal hemorrhage | 24 (-6/+24) hours
  parenchymal hemorrhage was defined as confluent bleeding occupying and causing mass effect
percentage of severe adverse events | 24 (-6/+24) hours
cerebral edema | 24 (-6/+24) hours
  cerebral edema was measured as the amount of midline shift of the brain on neuroimaging
death due to all causes | Day 7 or during hospitalization
occurrence rate of the distal emboli after first pass | immediately after first pass
  The emboli means occlusion of the distal artery determined by DSA.
occurrence rate of extracranial hemorrhage | 24 (-6/+24) hours
  extracranial hemorrhage means other bleeding events except intracranial hemorrhage

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: Undecided